CLINICAL TRIAL: NCT00959738
Title: A Prospective Multicenter Randomized Controlled Clinical Trial to Compare the Method of Protective Diverting Loop Ileostomy With or Without the Support of a Plastic Rod
Brief Title: Diverting Loop Ileostomy: With or Without Rod
Acronym: ROLLI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difference found in interim analysis, not ethical to continue
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Lukas Bruegger MD, Bern University Hospital, Department of Visceral Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 061/08
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Ileostomy; Rectal Neoplasms
Keywords: loop ileostomy; quality of life; morbidity; Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): diverting loop ileostomy with rod
  Interventions: Procedure: Diverting loop ileostomy with rod
- B (Other): diverting loop ileostomy without rod
  Interventions: Procedure: diverting loop ileostomy without rod

INTERVENTIONS:
Procedure: Diverting loop ileostomy with rod — Diverting loop ileostomy with rod
  Arms: A
Procedure: diverting loop ileostomy without rod — diverting loop ileostomy without rod
  Arms: B

SUMMARY:
Diverting ileostomies are created to protect a rectal anastomosis or in situations with a risk of intestinal perforation. Currently, the application of a rod to hinder slippage of the loop is an established technique to perform a diverting loop ileostomy. However, various "rod-less" techniques have been described and are performed with similar success. The aim of this study is to determine, whether a modification (without rod) of the current standard method of protective loop ileostomy formation (with rod) could improve ileostomy specific morbidity. Secondary endpoints include stoma care, determinants of quality of life and stoma function.

DETAILED DESCRIPTION:
Background

For rectal anastomoses within 6 cm of the anal verge, leakage rates are up to 15%. Here liberal use of protective stomas is widely accepted. Fecal diversion by loop ostomy may also be performed after extended adhesiolysis with serosal lesions and risk of intestinal perforation, in patients with obstructing rectal tumours requiring neoadjuvant radio-chemotherapy or in patients with complex anorectal injuries or fistulas. Generally, diverting loop ileostomies are secured at skin level by means of a supporting device in order to prevent retraction of the loop ileostomy into the abdomen. Nevertheless, due to the supporting rod, difficulties may occur in applying a stoma bag correctly and leakage of feces onto the skin may occur even with correct eversion of the afferent limb. Despite easier application of stoma bags and therefore reduced risk of skin irritation, none of these alternative techniques are established. In various non-randomized studies rodless loop ileostomies were described with an overall morbidity between 3 and 39%. However definition of morbidity varies significantly in these studies and randomised controlled trials are missing so far.

Objective

The aim of this study is to determine, whether a modification (without rod) of the current standard method of protective loop ileostomy formation (with rod) could improve ileostomy specific morbidity. Secondary endpoints include stoma care, determinants of quality of life and stoma function.

Methods

The study is designed as multi-institutional, randomized controlled, two-armed study. Patients scheduled for a protective loop ileostomy and meeting the eligibility criteria will be randomized to creation of a loop ileostomy with or without sustaining rod.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for planned protective loop ileostomy

Exclusion Criteria

* patients with long-term use of corticosteroids (> 15 mg prednisolone equivalent)
* immunosuppressive agent rapamune

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Severe stoma specific morbidity rate | postoperative during 2 weeks, 3 months postoperative

SECONDARY OUTCOMES:
Rate of patients reaching self-sufficient stoma care | postoperative during 2 weeks
Time used by the stoma nurses for instructing and assisting patients | preoperative, 2 weeks and 3 months postoperative
  Measured in total hours from the intervention up to 3 months postoperatively
Quality of life (QoL) by a stoma quality of life scale | postoperative during 2 weeks, 3 months postoperative
Predictive factors for stomal complications | postoperative during 2 weeks, 3 months postoperative

OTHER OUTCOMES:
Length of hospital stay, measured in days after intervention | postoperative during 2 weeks, 3 months postoperative
Change in eversion of the stoma nipple at postoperative days 2, 4, 6, 8, 14, 30, 60, 90 | postoperative days 2, 4, 6, 8, 14, 30, 60, 90
Start of stomal activity in hours after intervention | postoperative during 2 weeks, 3 months postoperative
Number of stoma bags and self-adhesive plates needed in the first month after the operation | postoperative during 2 weeks, 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Lukas E Bruegger, MD, Principal Investigator — Bern University Hospital,Dep. of Visceral and Transplant Surgery Switzerland
Locations (1):
- Bern University Hospital, Dep. of Visceral and Transplant Surgery, Bern, Switzerland

REFERENCES:
- [Background] Rosen HR, Schiessel R. [Loop enterostomy]. Chirurg. 1999 Jun;70(6):650-5. doi: 10.1007/s001040050701. German. PMID 10427451
- [Background] Gastinger I, Marusch F, Steinert R, Wolff S, Koeckerling F, Lippert H; Working Group 'Colon/Rectum Carcinoma'. Protective defunctioning stoma in low anterior resection for rectal carcinoma. Br J Surg. 2005 Sep;92(9):1137-42. doi: 10.1002/bjs.5045. PMID 15997447
- [Background] Moran B, Heald R. Anastomotic leakage after colorectal anastomosis. Semin Surg Oncol. 2000 Apr-May;18(3):244-8. doi: 10.1002/(sici)1098-2388(200004/05)18:33.0.co;2-6. PMID 10757890
- [Background] Karanjia ND, Corder AP, Bearn P, Heald RJ. Leakage from stapled low anastomosis after total mesorectal excision for carcinoma of the rectum. Br J Surg. 1994 Aug;81(8):1224-6. doi: 10.1002/bjs.1800810850. PMID 7953369
- [Background] Silva MA, Ratnayake G, Deen KI. Quality of life of stoma patients: temporary ileostomy versus colostomy. World J Surg. 2003 Apr;27(4):421-4. doi: 10.1007/s00268-002-6699-4. PMID 12658485
- [Background] Amin SN, Memon MA, Armitage NC, Scholefield JH. Defunctioning loop ileostomy and stapled side-to-side closure has low morbidity. Ann R Coll Surg Engl. 2001 Jul;83(4):246-9. PMID 11518371
- [Background] Edwards DP, Leppington-Clarke A, Sexton R, Heald RJ, Moran BJ. Stoma-related complications are more frequent after transverse colostomy than loop ileostomy: a prospective randomized clinical trial. Br J Surg. 2001 Mar;88(3):360-3. doi: 10.1046/j.1365-2168.2001.01727.x. PMID 11260099
- [Background] Bada-Yllan O, Garcia-Osogobio S, Zarate X, Velasco L, Hoyos-Tello CM, Takahashi T. [Morbi-mortality related to ileostomy and colostomy closure]. Rev Invest Clin. 2006 Nov-Dec;58(6):555-60. Spanish. PMID 17432286
- [Background] Goldstein ET, Williamson PR. A more functional loop ileostomy rod. Dis Colon Rectum. 1993 Mar;36(3):297-8. doi: 10.1007/BF02053516. PMID 8449139
- [Background] Unti JA, Abcarian H, Pearl RK, Orsay CP, Nelson RL, Prasad ML, Duarte B, Leff MM, Tan AB. Rodless end-loop stomas. Seven-year experience. Dis Colon Rectum. 1991 Nov;34(11):999-1004. doi: 10.1007/BF02049964. PMID 1935478